CLINICAL TRIAL: NCT05411276
Title: A Real-World Study of Pyrotinib Maleate in the Treatment of Advanced/Metastatic Non-Small Cell Lung Cancer With Rare Mutations in HER2
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Beijing Chest Hospital (Other)
Collaborators: Jiangsu HengRui Medicine Co., Ltd. (Industry)
Responsible Party: Principal Investigator, Ying Hu, Director of the Second Department of Oncology, Beijing Chest Hospital
Other Study IDs: KY-2021-012
Record Dates: First submitted 2022-06-06; First posted 2022-06-09 (Actual); Last update posted 2022-06-09 (Actual); Status verified 2022-06

CONDITIONS: HER2 Mutant Non-small Cell Lung Cancer
Keywords: Non-Small Cell Lung Cancer; Rare Mutation of HER2; Pyrotinib
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Year
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Group 1: HER2 rare mutation advanced/metastatic non-small lung cancer (IV)
  Interventions: Drug: Pyrotinib maleate

INTERVENTIONS:
Drug: Pyrotinib maleate — Pyrotinib maleate tablets 400 mg/day, oral within 30 minutes after breakfast, every 4 weeks is a cycle

SUMMARY:
At present, the main characteristics of the enrolled population in the clinical study of HER2-mutated non-small cell lung cancer are the YVMA mutation type. There are no relevant clinical trials specifically targeting rare mutation types. Pyrotinib has been approved for the treatment of HER2-positive advanced breast cancer in China, and pyrotinib has shown good development prospects in the treatment of advanced non-small cell lung cancer. The purpose of this study is to observe the efficacy and safety of pyrotinib maleate in patients with HER2 rare mutation in advanced non-small cell lung cancer.

ELIGIBILITY:
Inclusion Criteria:

* 1. Age: 18-70 years old;
* 2. Advanced/metastatic non-small lung cancer (IV) confirmed by pathology with measurable lesions;
* 3. HER2 mutation and amplification confirmed by gene testing of tumor tissue or blood, pleural effusion, cerebrospinal fluid and other specimens;
* 4. ECOG：0-1;
* 5. At least one radiographically measurable lesion
* 6. Expected survival period ≥ 3 months
* 7. Left ventricular ejection fraction (LVEF) ≥ 50% on echocardiography
* 8. Before using the drug for the first time, it was confirmed by laboratory tests that the subject's bone marrow function, liver and kidney function met the following requirements：

  1. Neutrophil count (ANC) ≥ 1,500/mm3 (1.5×109/L);
  2. Platelet count (PLT) ≥ 100,000/mm3 (100×109/L);
  3. Hemoglobin (Hb) ≥ 8 g/dL (80 g/L);
  4. Serum creatinine (SCr) ≤ 1.5 times the upper limit of normal (ULN) or creatinine clearance ≥ 60 ml/min;
  5. Total bilirubin (TBIL) ≤ 1.5 times the upper limit of normal (ULN);
  6. Aspartate aminotransferase (AST) or alanine aminotransferase (ALT) levels ≤ 2.5 times the upper limit of normal (ULN), and subjects with liver metastases should be ≤ 5×ULN;
  7. International normalized ratio (INR) ≤ 1.5, prothrombin time (PT) and activated partial thromboplastin time (APTT) ≤ 1.5 times ULN;
  8. Urine protein <2+; if urine protein ≥2+, the 24-hour urine protein quantification shows that protein must be ≤1g;
* 9. The medication regimen of the subjects during the clinical diagnosis and treatment was pyrotinib as a single drug
* 10. Patients voluntarily entered the study and signed informed consent form (ICF)

Exclusion Criteria:

* Common types of HER2 mutations: YVMA mutations;
* Patients with hypertension that cannot be well controlled by antihypertensive drug treatment (systolic blood pressure>140 mmHg, diastolic blood pressure>90 mmHg); Uncontrolled or severe cardiovascular disease, such as refractory angina pectoris, congestive heart failure occurred within 6 months before screening; Myocardial infarction within 12 months prior to screening; Any history of clinically significant ventricular arrhythmia, prolonged QT interval; History of cerebrovascular accident, symptomatic coronary heart disease requiring drug treatment;
* There are significant digestive tract dysfunction, which may affect the intake, transport or absorption of oral drugs (such as inability to swallow, chronic diarrhea, intestinal obstruction, etc.);
* Subjects with a recent history of active bleeding, clinically significant bleeding symptoms, and a clear bleeding tendency, such as hemoptysis, gastrointestinal bleeding, hemorrhagic gastric ulcer, positive fecal occult blood at baseline and above, etc.;
* Major surgical operations or severe traumatic injuries, fractures, or poorly healing wounds have been received within 4 weeks;
* Uncontrollable history of important respiratory system such as bronchiectasis, chronic obstructive pulmonary disease, lung abscess, pulmonary embolism, etc.;
* Active serious clinical infection (>NCI-CTCAE, 5.0 version 2 infection standard) and viral infections such as hepatitis B, hepatitis C, syphilis and HIV;
* Symptomatic brain metastases or meningeal metastases;
* Combined with previously untreated tumors other than primary lung cancer;
* Participated in clinical trials of other drugs within 4 weeks before the start of the study;
* Received treatment with pyrotinib maleate;
* Those who have serious adverse reactions and allergies to pyrotinib maleate;
* Pregnant or lactating female subjects, female subjects who are fertile and have a positive baseline pregnancy test, or subjects of childbearing age who are unwilling to take effective contraceptive measures throughout the trial;
* Have serious concomitant diseases, or any other conditions that the investigator considers unsuitable to participate in this study.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: HER2 rare mutation advanced/metastatic non-small lung cancer (IV)
Sampling Method: Non-Probability Sample
Enrollment: 15 (Estimated)
Dates: Start 2022-06-30 (Estimated); Primary Completion 2023-12-31 (Estimated); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
ORR | 2 Year
  It is defined as the proportion of patients whose tumors shrink to a predetermined size and maintain a minimum time limit. It includes the cases of CR and PR.

SECONDARY OUTCOMES:
PFS | 1 Year
  From the date Into this study to tumor progression or death for any
OS | 2 Year
  The time from the beginning of treatment to the death of the subject due to various reasons, calculated by the intended treatment population (ITT)
DCR | 2 Year
  the rate of CR, PR plus SD
AEs and SAEs | 1 Year
  Number of Participants With adverse events (AEs) and serious adverse events (SAEs) Incidence, nature, and severity of adverse events graded according to the NCI CTCAE v5.0.
QoL | 1 Year
  The quality of life of the subjects was assessed according to the EORTC QLQ-C30 quality of life questionnaire.

CONTACTS AND LOCATIONS:
Overall Officials: Ying Hu, Doctor, Principal Investigator — Beijing Chest Hospital